CLINICAL TRIAL: NCT02901314
Title: My Recordable On-Demand Audio Discharge Instructions (MyROAD)
Brief Title: My Recordable On-Demand Audio Discharge Instructions
Acronym: MyROAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Greetings (Unknown)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Associate Chief Nursing officer, Nursing Research and Innovation, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-122
Record Dates: First submitted 2016-09-01; First posted 2016-09-15 (Estimated); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: usual care education versus education with a pre-recorded card with heart failure instructions
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyRoad (Experimental): Receives usual care heart failure education before discharge AND a card at discharge that provided pre-recorded audio messages that can be played back on-demand on 4 themes: heart failure signs/symptoms assessment, medications, activity and exercise and diet and a general message about the importance of follow-up post discharge and following the plan of care.
  Interventions: Other: on-demand audio messages of heart failure education themes
- Usual care (No Intervention): Receives usual care heart failure education before discharge

INTERVENTIONS:
Other: on-demand audio messages of heart failure education themes
  Arms: MyRoad

SUMMARY:
Non-adherence to the heart failure (HF) plan of care after hospital discharge has been associated with clinical outcomes, including the combined endpoint of all-cause mortality and rehospitalization for decompensated HF. Patients and informal caregivers receive education materials but may not act due to multiple factors. A recorded message that could be repeatedly played by patients and caregivers might increase adherence to post-discharge self-care behaviors and early follow-up appointments, and have clinical benefits related to a reduction in all-cause mortality and rehospitalization. The purposes of this randomized, controlled study are to examine the effects of use of a novel MyROAD (Recordable On-Demand Audio Discharge) card, given to patients at discharge. The aims of this single-blind, placebo-controlled study are to examine the effects of recorded messages that can be replayed post discharge (delivered via the MyROAD card) on multiple subjective and objective clinical outcomes.

DETAILED DESCRIPTION:
Non-adherence to the heart failure (HF) plan of care after hospital discharge has been associated with clinical outcomes, including the combined endpoint of all-cause mortality and rehospitalization for decompensated heart failure. Most patients are discharged with a complex set of instructions that include multiple medications (and differing mediation administration plans), sodium restricted diet, fluid management actions (daily weight monitoring and in some cases, fluid restriction), monitoring signs and symptoms of HF, activity and exercise, and when to return for follow-up. At discharge, patients (and their families) may not understand that heart failure is chronic. Improvement in quality of life may be dependent on patients' acceptance of HF as a chronic, irreversible condition that requires self-care monitoring and behaviors (for example, becoming or staying physically active), even when they feel fine. To decrease the complexity of understanding heart failure, patients receive a heart failure handbook and a "zones" 1-page handout before discharge. In addition, they can watch multiple video clips of many heart failure topics and discuss heart failure self-care with the hospital healthcare team. However, patients may not read (or view) education materials due to health literacy issues, cognitive decline, eyesight issues, fatigue, or depression. Patients may rely on lay (family) caregivers to understand self-car expectations and be active partners in care. Caregivers engaged in patients' care may not be present at discharge or may have preconceived or inaccurate ideas about heart failure self-care after discharge. A recorded message that could be repeatedly played by patients and caregivers might increase adherence to post-discharge self-care behaviors and 7-day follow-up appointments, and have clinical benefits related to a reduction in all-cause mortality and rehospitalization. The purpose of this randomized, controlled study are to examine the effects of use of a novel MyROAD (Recordable On-Demand Audio Discharge) card, given to patients at discharge. The aims of this single-blind, placebo-controlled study are to examine the effects of recorded messages that can be replayed post discharge (delivered via the MyROAD card) on (1) 45-, 90-, and 180-day first occurrence and (2) time to first occurrence of all-cause and HF-related hospitalization, emergency department visits and death/ cardiac transplantation/ventricular assist device, (3) 45-day quality of life (Kansas City Cardiomyopathy Questionnaire), symptoms (investigator initiated tool; used in previous research), functional status (Duke Activity Status Index) and perceived adherence to activity recommendations (investigator initiated tool; used in previous research), and (4) 7-day follow-up appointment with the healthcare provider assigned before discharge. A total of 1066 patients (968 + 10% attrition) with decompensated heart failure will be randomized to either usual care or usual care and receiving a MyROAD card at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Not referred for cardiac transplantation or ventricular assist device during the index hospitalization,
* Minimum age 18 years (no upper age limit),
* Ability to read and write,
* Discharge to home or to a family member's home and has control of making self-care decisions,
* Willing to participate; which requires three (3) follow-up telephone calls post-discharge.

Exclusion Criteria:

* Chart documented psychiatric or cognitive conditions that limit ability to understand or adhere to self-care recommendations (Alzheimer's condition, dementia, schizophrenia, other neurological history that impairs memory),
* Plans to discharge to assisted living apartment/center, skilled nursing facility or hospice care center,
* Receiving home hospice or palliative care; or has a medical condition reflecting less than 1 year of survival (cachexia, end stage liver disease or cancer or non-ambulatory New York Heart Association functional class IV heart failure),
* Post-cardiac transplantation or ventricular assist device placement,
* Currently enrolled in another experimental heart failure research study,
* Chronic renal failure and receiving chronic hemodialysis therapy for an estimated glomerular filtration rate < 30 mL/minute/1.73 m2,
* A non-traditional form of heart failure (hypertrophic or restrictive forms of cardiomyopathy, congenital heart disease or Takotsubo cardiomyopathy).
* Wheelchair bound, uses a cane or walker, or unable to carry out physical activity, including walking,due to a chronic disability or documented medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2487 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Cleveland Clinic main campus, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Hillcrest hospital, Mayfield Heights, Ohio
  - Cleveland Clinic Medina Hospital, Medina, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with decompensated heart failure HF with preserved or reduced ejection fraction when hospitalized and New York Heart Association FC III or ambulatory IV. Dates of enrollment occurred between March 2016 to June 2019.
Pre-assignment Details: Of the 2487 patients enrolled, 1073 met inclusion criteria and were randomized to either usual care or usual care + intervention (My Recordable On-Demand Audio Discharge Instructions MyROAD card).
Groups:
- MyRoad: Receives usual care heart failure education before discharge AND a card at discharge that provided pre-recorded audio messages that can be played back on-demand on 4 themes: heart failure signs/symptoms assessment, medications, activity and exercise and diet and a general message about the importance of follow-up post discharge and following the plan of care.
  on-demand audio messages of heart failure education themes
Period: Overall Study
Arm/Group | MyRoad | Usual Care
Started | 538 | 535
Completed | 506 | 491
Not Completed | 32 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyRoad | Usual Care | Total
Number analyzed (Participants) | 506 | 491 | 997
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (11.2) | 73.1 (11.0) | 72.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 206 | 412
  Male | 300 | 285 | 585
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 123 | 120 | 243
  White | 375 | 362 | 737
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 506 | 491 | 997
Marital status [Count of Participants; unit: Participants]
  Single | 66 | 75 | 141
  Married | 255 | 239 | 494
  Divorced/Separated | 66 | 67 | 133
  Widowed | 108 | 104 | 212
  Co-habitate (living with partner) | 11 | 6 | 17
Location [Count of Participants; unit: Participants]
  Main campus | 288 | 282 | 570
  Hillcrest | 115 | 116 | 231
  Fairview | 73 | 66 | 139
  Medina | 30 | 27 | 57
Do you currently live with another person? [Count of Participants; unit: Participants]
  Yes | 390 | 374 | 764
  No | 116 | 117 | 233
Do you have someone to confide in? [Count of Participants; unit: Participants]
  Yes | 492 | 482 | 974
  No | 13 | 9 | 22
  Missing survey response | 1 | 0 | 1
Highest level of education completed [Count of Participants; unit: Participants]
  Less than high school graduate | 75 | 69 | 144
  General Educational Development (GED) | 8 | 9 | 17
  High school graduate | 182 | 172 | 354
  Some college or professional training post high school | 131 | 143 | 274
  Associate degree | 17 | 20 | 37
  Bachelor's degree | 61 | 47 | 108
  Master's degree | 24 | 18 | 42
  Doctoral degree | 8 | 13 | 21
Employment status [Count of Participants; unit: Participants]
  Employed full or part-time | 60 | 61 | 121
  Unemployed by choice | 22 | 11 | 33
  Sick leave or disability | 46 | 57 | 103
  Retired due to HF | 60 | 51 | 111
  Retired, not due to HF | 318 | 310 | 628
  Other | 0 | 1 | 1
Consider how well you live on income [Count of Participants; unit: Participants]
  Comfortable, more than enough | 158 | 137 | 295
  Have enough to make ends meet | 224 | 232 | 456
  Do not have enough to make ends meet | 124 | 122 | 246
In general, would you say your health is [Count of Participants; unit: Participants]
  Poor | 135 | 119 | 254
  Fair | 200 | 222 | 422
  Good | 138 | 110 | 248
  Very good | 23 | 29 | 52
  Excellent | 10 | 11 | 21
Health care services [Count of Participants; unit: Participants]
  When was the last time you were in hospital for any reason?: Left the hospital within the last 7 days | 33 | 34 | 67
  When was the last time you were in hospital for any reason?: Left the hospital 2 weeks ago (8-14 days ago) | 50 | 40 | 90
  When was the last time you were in hospital for any reason?: Left the hospital 3-4 weeks ago (15-30 days ago) | 59 | 43 | 102
  When was the last time you were in hospital for any reason?: Left the hospital over 1 month ago but <3 months ago | 125 | 126 | 251
  When was the last time you were in hospital for any reason?: Longer than 3 months ago | 239 | 248 | 487
  When was the last time you were in hospital for any reason?: Don't remember or never been in hospital | 0 | 0 | 0
  When was the last time you were hospitalized for heart failure?: Left the hospital within the last 7 days | 28 | 29 | 57
  When was the last time you were hospitalized for heart failure?: Left the hospital 2 weeks ago (8-14 days ago) | 36 | 32 | 68
  When was the last time you were hospitalized for heart failure?: Left the hospital 3-4 weeks ago (15-30 days ago) | 50 | 36 | 86
  When was the last time you were hospitalized for heart failure?: Left the hospital over 1 month ago but <3 months ago | 90 | 97 | 187
  When was the last time you were hospitalized for heart failure?: Longer than 3 months ago | 300 | 292 | 592
  When was the last time you were hospitalized for heart failure?: Don't remember or never been in hospital | 2 | 5 | 7
  When was last time you were in hospital for your heart, but not heart failure: Left the hospital within the last 7 days | 15 | 12 | 27
  When was last time you were in hospital for your heart, but not heart failure: Left the hospital 2 weeks ago (8-14 days ago) | 24 | 15 | 39
  When was last time you were in hospital for your heart, but not heart failure: Left the hospital 3-4 weeks ago (15-30 days ago) | 27 | 21 | 48
  When was last time you were in hospital for your heart, but not heart failure: Left the hospital over 1 month ago but <3 months ago | 78 | 85 | 163
  When was last time you were in hospital for your heart, but not heart failure: Longer than 3 months ago | 352 | 346 | 698
  When was last time you were in hospital for your heart, but not heart failure: Don't remember or never been in hospital | 10 | 12 | 22
Heart failure etiology [Count of Participants; unit: Participants]
  Ischemic | 265 | 259 | 524
  Idiopathic | 97 | 101 | 198
  Hypertensive | 49 | 42 | 91
  Valvular heart disease | 82 | 77 | 159
  Alcoholic | 7 | 3 | 10
  Postpardum | 1 | 0 | 1
  Chemotherapy | 2 | 7 | 9
  Other | 3 | 2 | 5
Ejection fraction % [Mean (Standard Deviation); unit: % of blood ejected with each contraction] | 41.3 (17.2) | 42.0 (16.8) | 41.6 (17.0)
Cardiac devices at admission or before hospital discharge [Count of Participants; unit: Participants]
  ICD (Implantable Cardioverter Defibrillator) | 88 | 84 | 172
  CRT (Cardiac Resynchronization Therapy) | 9 | 6 | 15
  CRT-D (Cardiac Resynchronization Therapy with Pacemaker) | 45 | 33 | 78
  DDD pacemaker (dual-chamber pacemaker) | 27 | 28 | 55
  AAI pacemaker (single chamber pacemaker operates in AAI mode) | 3 | 2 | 5
  None | 332 | 333 | 665
  Other | 2 | 5 | 7
Drug classes at discharge [Count of Participants; unit: Participants]
  Angiotensin-converting enzyne inhibitors (ACE-i) | 145 | 117 | 262
  Angiotensin receptor neprilysin inhibitor (ARNI) | 29 | 15 | 44
  Angiotensin receptor blocker (ARB) | 67 | 58 | 125
  Beta blocker | 398 | 401 | 799
  Aldosterone antagonist | 136 | 129 | 265
  Sinus node funny channel inhibitor | 1 | 0 | 1
  Statin | 321 | 328 | 649
  Hydralazine | 87 | 103 | 190
  Nitrate | 150 | 171 | 321
  Digoxin | 77 | 68 | 145
  Loop diuretic | 457 | 449 | 906
  Thiazide or Thiazide like diuretic | 15 | 28 | 43
Charlson Comorbidity Index [Count of Participants; unit: Participants] — The Charlson Comorbidity Index (CCI) is a measurement tool to predict mortality risk based on the number and severity of co-morbidities.
  Minimum score 0 Maximum score 28
  A score of zero indicates no risk and the highest score indicates a higher risk of mortality.
  Participants
    >1.5 but <2.5 | 193 | 163 | 356
    >2.5 but <3.5 | 140 | 161 | 301
    >3.5 but <4.5 | 97 | 86 | 183
    >4.5 but <6.5 | 65 | 65 | 130
    >6.5 | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Rehospitalized With Heart Failure
Description: Number of patients re-hospitalized with heart failure.
Time Frame: 30 day
Population: Some patients were not included in the 30 day data due to heart failure related death, LVAD, or heart transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 496 | 475
Participants
  Rehospitalized | 71 | 78
  Not rehospitalized | 425 | 397

2. Secondary Outcome: Number of Patients Scheduled for 7-day Follow-up Appointment With the Healthcare Provider Before Discharge
Description: Adherence to 7-day follow-up appointment with a healthcare provider; by medical record chart review
Time Frame: Discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 506 | 491
Participants | 290 | 285

3. Secondary Outcome: Quality of Life (Health Status)
Description: Quality of life was measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is a 23-item questionnaire that measures physical limitations, symptoms, self-efficacy, social interference and quality of life. The KCCQ is a standardized score from 0 to 100 points. A score of 0 is the lowest quality of life (poor) and score of 100 is the highest quality of life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 506 | 491
score on a scale | 46.1 (17.0) | 45.5 (17.3)

4. Secondary Outcome: Quality of Life (Health Status)
Description: as for outcome 3
Time Frame: 45 day
Population: The number analyzed in both groups was lower than the number enrolled due to being unable to reach patients by phone for follow-up or the patient was deceased.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 470 | 433
score on a scale | 62.6 (21.4) | 64.5 (22.5)

5. Secondary Outcome: Symptoms
Description: 29-item list of heart failure-related symptoms. Patients were asked to consider any symptoms they experienced in the last 2 weeks and choose all that apply. Patients could also check "do not weigh self" and "no signs or symptoms of anything abnormal". The median [Q1, Q3] number of symptoms was reported between groups.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: Symptoms
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 506 | 491
Symptoms | 8.0 [5.0 to 11.0] | 8.0 [5.00 to 11.0]

6. Secondary Outcome: Symptoms
Description: as for outcome 5
Time Frame: 45 days
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Symptoms
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 471 | 434
Symptoms | 4.0 [2.0 to 6.0] | 4.0 [1.0 to 6.0]

7. Secondary Outcome: Functional Status
Description: Duke Activity Status Index (DASI) is a 12-item questionnaire using Likert scale that determines a patient's ability to participate in common, everyday activities without difficulty including self-care activities (e.g., ambulation, housework, yard work, sexual relations, and recreational activities. This is a patient-reported tool that measures functional status in patients with heart failure.
  Scores range from 0 (no functional capacity = worst score) to 58.2 (highest functional capacity = best score).
Time Frame: Baseline
Population: Patients enrolled in the study were later excluded (e.g., due to death, discharged to Skilled Nursing Facility, dialysis, or left ventricular assist device).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 506 | 491
score on a scale | 19.7 (11.1) | 19.0 (10.6)

8. Secondary Outcome: Functional Status
Description: Duke Activity Status Index (DASI) is a 12-item questionnaire. This is a patient-reported tool that measures functional status in patients with heart failure. Patients were called by telephone and asked to rate their ability to do daily activities (e.g., personal care, ambulation, household tasks, sexual function, and recreation).
  Scores range from 0 (no functional capacity = worst score) to 58.2 (highest functional capacity = best score).
Time Frame: 45 day
Population: The number analyzed in both groups was lower than the number enrolled due to being unable to reach patients by phone or the patient was deceased (medical record chart review).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 470 | 433
score on a scale | 18.1 (10.5) | 18.3 (10.8)

9. Secondary Outcome: Adherence to Activity Recommendations
Description: Modified PACE tool; used in previous research. Patients were asked to self-report their perceived adherence to activity recommendations by selecting the option on a checklist that matched their activity level.
Time Frame: Baseline
Population: Patients enrolled in the study were later excluded (e.g., due to death, discharged to a Skilled Nursing Facility, dialysis, or left ventricular assist device).
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 467 | 433
Participants
  I do not walk now | 164 | 165
  I've been thinking of starting | 207 | 176
  Walk 2/week <10 minutes | 17 | 14
  Walk 2/week >10 minutes | 12 | 16
  Walk 3-5 days/week <10 minutes | 7 | 11
  Walk 3-5 days/week for 10-20 minutes | 15 | 6
  Walk 3-5 days/week >20 minutes | 7 | 12
  Walk 6-7 days/week <10 minutes | 2 | 3
  Walk 6-7 days/week for 10-20 minutes | 7 | 8
  Walk 6-7 days/week >20 minutes | 6 | 4
  Began moderate or vigorous exercise <3 x week | 5 | 3
  Moderate exercise 3+ per week the last 1-6 months | 6 | 8
  Moderate exercise 3+ week for 7 months | 8 | 6
  Vigorous exercise 3-5 week for 1-6 months | 1 | 1
  Vigorous exercise 3-5 week >12 months | 2 | 0

10. Secondary Outcome: Adherence to Activity Recommendations
Description: Modified PACE tool; used in previous research. Patient's were contacted by telephone and asked to self-report their perceived adherence to activity recommendations.
Time Frame: 45 day
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 467 | 433
Participants
  I do not walk now | 186 | 161
  I've been thinking of starting | 162 | 148
  Walk 2/week <10 minutes | 8 | 7
  Walk 2/week >10 minutes | 12 | 11
  Walk 3-5 days/week <10 minutes | 15 | 17
  Walk 3-5 days/week for 10-20 minutes | 20 | 14
  Walk 3-5 days/week >20 minutes | 6 | 11
  Walk 6-7 days/week <10 minutes | 11 | 10
  Walk 6-7 days/week for 10-20 minutes | 10 | 20
  Walk 6-7 days/week >20 minutes | 10 | 8
  Began moderate or vigorous exercise <3 x week | 10 | 8
  Moderate exercise 3+ per week the last 1-6 months | 12 | 14
  Moderate exercise 3+ week for 7 months | 3 | 4
  Vigorous exercise 3-5 week for 1-6 months | 1 | 0
  Vigorous exercise 3-5 week >12 months | 1 | 0

11. Secondary Outcome: Number of All-cause Re-hospitalization, Death, Left Ventricular Assist Device (LVAD), Cardiac Transplant (Composite Outcome)
Description: All-cause re-hospitalization, death, left ventricular assist device (LVAD), or cardiac transplant via medical record chart review; interview (telephone call).
Time Frame: 90 days
Population: The number analyzed in both groups was lower than the number enrolled due to being unable to locate information in the medical record or the patient was deceased.
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 503 | 488
Participants | 243 | 262

12. Secondary Outcome: Number of All-cause Re-hospitalization, Death, Left Ventricular Assist Device (LVAD), Cardiac Transplant (Composite Outcome)
Description: as for outcome 11
Time Frame: 180 days
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 497 | 483
Participants | 331 | 322

13. Secondary Outcome: Number of Patients Rehospitalized With Heart Failure
Description: Number of patients rehospitalized with heart failure via chart review; interview (telephone call).
Time Frame: 45 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 485 | 465
Participants | 91 | 104

14. Secondary Outcome: Number of Patients Rehospitalized With Heart Failure
Description: Number of patients rehospitalized with heart failure via chart review
Time Frame: 90 days
Population: The number analyzed in both groups was lower than the number enrolled due to being unable to locate information in the medical record chart.
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 458 | 440
Participants | 135 | 138

15. Secondary Outcome: Number of Patients Rehospitalized With Heart Failure
Description: Number of patients rehospitalized with heart failure via chart review; interview (telephone call).
Time Frame: 180 days
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 421 | 400
participants | 192 | 183

16. Secondary Outcome: Number of Patients With All-cause Rehospitalization, Death or Emergency Department Visit
Description: Number of patients with all-cause rehospitalization, death, or emergency department visits within 180 days. Information is obtained via medical record chart review.
Time Frame: 180 days
Population: patients enrolled and discharged from the hospital alive; that we were able to obtain 180 day data on, assessed treatment group compared to usual care group
Measure: Count of Participants; unit: Participants
Arm/Group | MyRoad | Usual Care
Number analyzed (Participants) | 497 | 483
Participants | 331 | 322

ADVERSE EVENTS:
Time Frame: Not applicable; the intervention was not directly related to patient events that could have occurred after receiving education; therefore no event data were collected
Description: For the 0 participants at risk (e.g., "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | MyRoad | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02901314/Prot_SAP_000.pdf